CLINICAL TRIAL: NCT03607929
Title: Effectiveness "HIDRATACION OPTIMA " During Labor in Reducing Time Dilation and Expulsion, Cesarean, Fever and Dehydration
Brief Title: HIDRATA Study: Efficacy of a Hydration Protocol in Nulliparous Women During Labor
Acronym: HYDRATA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Ana Belén Hernández López, Midwife, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PuertadeHierro; PI15/00897 (Other Grant/Funding Number: Ministry of Health of Spain)
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Labor Long; Nulliparity; Premature Rupture of Membrane; Pregnancy, Prolonged; Pregnancy
Keywords: ARE; deshydration; adverse events; cesarean; fever
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Pregnancy, Prolonged; Fever | interventions — Optimal Pressed Ceramic; Control Groups

STUDY DESIGN:
Intervention Model Description: INTERVENTION GROUP " OPTIMAL HYDRATION" LABOR: they will be initiated the administration of crystalloid solutions in continuous perfusion at a rate of 200ml/h, until delivery, alternating each of them: (1)Physiological Serum (2)Physiological Serum (3)Ringer Lactate. The oral intake of mineral water will be promoted, at a rate of 100ml/h. To avoid bias, the mineral water will be administered by the research team.
  IMMEDIATE PUERPERIUM: Women who have had a low-risk delivery will drink mineral water at a rate of 100ml / h during the two hours of the immediate puerperium. Suspending Hydration i.v.
  CONTROL GROUP " VARIABILITY IN HYDRATION" The women will be hydrated in accordance with the midwives' experience, training and clinical criteria, either independently or jointly with the attending clinicians (obstetricians, gynecologists and anesthetists).
Who Masked: Participant, Outcomes Assessor
Masking Description: The methodology for carrying out the clinical trial followed the directives proposed in the CONSORT 2010 Statement: Updated guidelines for reporting parallel group randomized trials (Schulz et al. 2010).
  Randomization and masking Women who fulfill the inclusion criteria will assigned in a masked manner into one of two groups according to a randomization list generated in the hospital's Care Research Unit using Epidat software version 3.1. Allocations will be disclosed through opaque, sealed, consecutively numbered envelopes at the moment the woman is recruited into the study . Given the difficulty of masking allocations from the persons carrying out the intervention and collecting the information, in addition to using objective variable measurement systems, collaborators will be blinded to the results during their analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- optimal and hydration (Experimental): Physiological Saline Solution 300 ml/h AND drink freely mineral water during labor
  Interventions: Procedure: optimal
- variability and hydration (Active Comparator): Other Solutions >o < 300 ml/h AND uncontrolled drink during labor
  Interventions: Procedure: variability

INTERVENTIONS:
Procedure: optimal — Physiological Saline Solution
  Other Names: controlled
  Arms: optimal and hydration
Procedure: variability — Other solutions
  Other Names: uncontrolled
  Arms: variability and hydration

SUMMARY:
Aim. To evaluate the efficacy of optimizing hydration during labor in nulliparous women with respect to reducing the duration of dilation and the second stage of labor, lowering the incidence of Cesarean sections and fever, and also with respect to changes in sodium and osmolarity in blood and urine, and 24 hour diuresis.

Background. In the international scientific community there is a lack of consensus regarding the most suitable hydration strategies to be used in the attention of nulliparous women during low risk birth. Insufficient hydration during labor is associated with increased maternal and neonatal morbidity.

Design. A randomized, controlled clinical trial with allocation concealment and masking during the evaluation of the results.

Methods. A study of nulliparous women whose births and newborn are attended in the Obstetric Service of a University Hospital. The women will be randomized to two groups: the "optimal hydration" group, that will be guaranteed 300 ml/h (intravenous crystalloids and water) with a minimum diuresis of 400 ml/24h; and the "variability in hydration" group, comprised of the administration of intravenous and clear liquid volumes, without any established perfusion rate, based on criteria established by the healthcare professional attending the birth, and without established minimum diuresis. Mother outcomes: duration of labor, Cesarean section, fever, dehydration. Newborn outcomes: distress, hypoglycemia, hyponatremia, jaundice, weight loss in 48h, breastfeeding difficulties. Analysis will be per-protocol. Statistical significance will be set at p<0.05 Discussion. The findings obtained in this study will provide new evidence for considering the benefits of providing women with suitable optimized hydration during labor. Diminishing the clinical practice variability related to hydration strategies applied to nulliparous women attended during labor through the use of a decision-making algorithm to administer optimal hydration, would imply improved health and safety for mothers and their newborn together with reduced maternal and neonatal morbidity.

Funding granted in 2015 by the Spanish Health Research Fund (PI 15/00897, Ministry of Health).

Keywords: hydration; dehydration; adverse events; labor; Cesarean section, fever.

DETAILED DESCRIPTION:
PRIMARY AIM:

To evaluate the efficacy of "optimal hydration" during labor in nulliparous pregnant women attended for spontaneous or induced deliveries with respect to the reduction in dilation times, second stage of labor and total labor time.

METHODOLOGY A randomized controlled clinical trial, with concealed allocation. The study is being carried out in a large university hospital belonging to the Spanish National Health System. The trial is being carried out in the Obstetrics Service in Hospital Universitario Puerta de Hierro Majadahonda, Madrid. All the study participants will be nulliparous women (women who have not given birth by the vaginal route), and their neonates, who are attended during either spontaneous labor (2-3 regular uterine contractions in 10 minutes, cervical effacement greater than 50% and 3-4 cm spontaneous dilatation) or induced labor (when labor is induced artificially). The sample size was estimated on the basis of cohorts previously studied by the same team of investigators in the same hospital which observed that women who had received liquid volumes of less than 300 ml/h during labor took a mean (SD) of 754 (251) minutes to complete the birth, whereas women who received a volume equal to or greater than 300 ml/h took a mean (SD) of 592 (287) minutes. Assuming a 95% confidence interval, in a bilateral contrast, with a statistical power of 90%, a population of 59 is required for each group. In addition, a 10% increase is taken into account for those lost to follow-up. Therefore, the final sample size is 130, with 65 women in each group.

Intervention group protocol: "optimal hydration" Women in this group will be attended by the 13 investigation team midwives who have agreed to collaborate with the study's clinical team. Attention will include: (A) administration of a volume of liquids equal to 300 ml/h during labor which is defined as from the moment of admittance to the delivery room until the birth of the child; (B) more than 80% of the volume will be perfused intravenously using a physiological saline solution; (C) the women will be encouraged to drink clear liquids from the moment of admittance to the delivery room until reaching 10 cm dilation, such liquids will only be bottled mineral water (80%) and isotonic drinks (20%); (D) the perfusion rate will be increased if the woman has diuresis lower than 400 ml in 24h or presents temperature equal to or greater than 37.8ºC.

Control group protocol: "variability in hydration" Women in this group will be attended by the 16 delivery room midwives who do not belong to the investigation team. The women will be hydrated in accordance with the midwives' experience, training and clinical criteria, either independently or jointly with the attending clinicians (obstetricians, gynecologists and anesthetists). The principal lines of attention will be: (A) administration of undetermined volumes of liquids during labor which is defined as from the moment of admittance to the delivery room until the birth of the child; (B) the volume will be perfused intravenously using physiological saline solution, Ringer's, 5% glucose, 10% glucose or voluven; (C) the women will be allowed to drink clear liquids at their own pace and to their liking from the moment of admittance to the delivery room until reaching 10 cm dilation, such liquids can be water and isotonic drinks; (D) changes in perfusion rate and diuresis or increases in temperature (higher then 37.7ºC) will not be evaluated.

Study procedures The midwife in the Obstetric Emergency department will verify whether women attending the service comply with the criteria for inclusion in the study but do not present any exclusion criteria. In such cases, the midwife will give the woman verbal and written information about the study. If the woman is willing to participate, she will have to return a signed Informed Consent form to the midwife. The woman will at this moment be assigned the next consecutive number for inclusion in the study. The midwife will open the corresponding envelope containing the information regarding the group to which the woman has been assigned. In the case of assignment to the "controled hydration" group, the midwife responsible for her attention will be one of the 13 in the investigating team. If the woman is assigned to the "uncontroled in hydration" group, the midwife responsible for her attention will be one of the 16 who do not belong to the investigating team.

Study measures

Maternal variables:

* Main Outcomes: duration of dilation, duration of second stage of labor, and total duration from onset of labor until the birth.
* Secondary Outcomes: times on oxytocin, with ruptured membrane and epidural anesthesia, incidence of Cesarean section, incidence of intrapartum fever (temperature equal to or higher than 38ºC) and postpartum fever, dehydration (diuresis lower than 400 ml in 24 h, osmolarity concentration in urine/blood, sodium in urine/blood), headaches, nausea, vomiting, confusional state, hyperglycemia (blood sugar higher than 120 mg/dl), difficulty establishing breastfeeding, badly controlled thirst, badly controlled pain.
* Sociodemographic variables: age, nationality, educational level.
* Clinical variables on admittance, intrapartum, immediate postpartum (first 2 hours) and intermediate postpartum period (24 and 48 hours).

Neonate variables:

* Neonate outcomes: distress, seizures, nausea, vomiting, tachypnea, hypoglycemia (glycemia lower than 40 ml/dl), hyponatremia (sodium in umbilical cord blood <130 mEq/L), fever (temperature equal to or higher than 38ºC), jaundice (requiring phototherapy), more than 7% weight loss in 48 h, difficulty initiating breast feeding.
* Variables related to the newborn child (from birth, at 24 and 48 h): ions (sodium, potassium and glucose) in umbilical cord blood, gender, weight (at birth, at 24 and 48 h), distress, temperature, desire to suckle, colostrum, initiation of breastfeeding, type of breastfeeding, jaundice and capillary bilirubin levels (24 and 48 h).

Data collection Information will be collected from: clinical histories, partogram, observation, physical examination, fetal monitoring, scales (adult and newborn), analytical values, vital signs, visual analogue scale for pain (from 0 to 10), sensation of nausea (from 0 to 5), sensation of thirst (from 0 to 10), Armstrong scale (dehydration evaluation), Bilitest (capillary bilirubin levels), Silverman test (respiratory distress at birth). Maternal laboratory values: antenatal and in the immediate postpartum. Requests for blood and urine samples and their extraction, together with all other analyses, will be carried out by the Emergency Obstetric Service midwife according to normal clinical practice. Neonate laboratory values: at the time of birth. Requests for analyses will be made by the midwife during the dilation phase. Taking advantage of the moment when other samples are taken according to normal clinical practice (umbilical cord pH and blood group), sample extractions will be carried out by the midwife or obstetrician attending the delivery. The midwife will be responsible for weighing the newborn in the delivery room and in the Obstetric Service ward. The variables corresponding to the immediate postpartum (24-48 h) will be recorded by ward nurses who will be blinded to the group assignments.

Data analysis Analyses will be carries by assigned treatment and by intention to treat. Mean differences will be presented for qualitative values, and relative risks, reductions of relative and absolute risk, and the number required to treat for qualitative variables. All variables will be shown with their 95% confidence interval. Statistical significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria: Women who:

* Are 18 years-of-age or older;
* With gestation between 37-41+3 weeks
* Have signed an informed consent form.

Exclusion Criteria: The following exclusion criteria will apply:

* Women who do not have sufficient understanding of the Spanish language or those with whom communication will be difficult
* Women with a multiple gestation
* Gestation with high maternal or neonatal risk
* Maternal pathology (metabolic diseases, preeclampsia, eclampsia, etc.)
* Fetal pathology
* Precipitated delivery; fetal death.

Criteria for leaving the study:

* Severe maternal complications during the immediate or intermediate postpartum periods that require admittance to the Intensive care Unit
* Neonatal complications that require admittance to the Neonatology Service for more than 48 hours
* If, once the study has started, the participant fails to cooperate during follow-up (delivery, during the immediate or intermediate postpartum periods) or decides to discontinue their participation.

Ages: 29 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
duration of labor | 24 hours
  total duration from onset of labor until the birth.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Belen Hernandez Lopez, Miswife, Principal Investigator — Midwife
Locations (1):
- Puerta de Hierro Majadahonda University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No